CLINICAL TRIAL: NCT03084640
Title: A Multicenter, Two Part, Phase 1B Study Evaluating Alternative Routes of Administration of CMP-001 in Combination With Pembrolizumab in Subjects With Advanced Melanoma
Brief Title: Phase 1B Study Evaluating Alternative Routes of Administration of CMP-001 in Combination With Pembrolizumab in Participants With Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-002
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose-Escalation - CMP-001 (SC) and Pembrolizumab (Experimental): Participants will receive up to 7 escalating dose levels (5 milligrams [mg], 7.5 mg, 10 mg, 12.5 mg, 15 mg, 17.5 mg, and 20 mg) of CMP-001 via SC injection once a week for 3 weeks and every 3 weeks thereafter until discontinuation of treatment in combination with pembrolizumab at its labelled dose and schedule.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab
- Part 1: Dose-Expansion - CMP-001 (SC) and Pembrolizumab (Experimental): Participants will receive RP2D (as determined in Part 1 dose-escalation phase) of CMP-001 via SC injection once a week for 3 weeks and every 3 weeks thereafter until discontinuation of treatment in combination with pembrolizumab at its labelled dose and schedule.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab
- Part 2: CMP-001 (SC and IT) and Pembrolizumab (Experimental): Participants will receive CMP-001 via SC injection once weekly for 2 weeks, then IT injection once weekly for 4 weeks, and SC injection once weekly for every 3 weeks thereafter until discontinuation of treatment in combination with pembrolizumab at its labelled dose and schedule. CMP-001 planned IT dose level in Part 2 will be up to 10 mg and the SC dose will be the RP2D determined from Part 1 dose-escalation phase of the study.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CMP-001 — CMP-001 will be administered SC as per the dose and schedule specified in the respective arms.
Drug: Pembrolizumab — Pembrolizumab will be administered as per the schedule specified in the respective arms.
  Other Names: Keytruda
Drug: CMP-001 — CMP-001 will be administered IT as per the dose and schedule specified in the respective arms.
  Arms: Part 2: CMP-001 (SC and IT) and Pembrolizumab

SUMMARY:
CMP-001-002 is a Phase 1b study of CMP-001 administered to participants with advanced melanoma who are either receiving pembrolizumab, or who have previously received an anti-programmed cell death protein 1 (anti-PD-1)/programmed death-ligand 1 (PD-L1) therapy for advanced melanoma, and who have not responded (that is, immunotherapy resistant).

This study will be conducted in two parts:

Part 1 will consist of a Dose Escalation Phase and a Dose Expansion Phase

* Dose Escalation Phase will be conducted to assess and identify a recommended phase 2 dose (RP2D) of CMP-001 for subcutaneous (SC) administration
* The Dose Expansion Phase is intended to further characterize the safety, pharmacodynamics, and preliminary evidence of antitumor activity of the RP2D of CMP-001 administered SC in combination with pembrolizumab

Part 2 will assess the safety and preliminary evidence of antitumor activity of CMP-001, administered both SC and intratumoral (IT) when given in combination with pembrolizumab.

Participants will continue treatment with CMP-001 in combination with pembrolizumab as long as they do not experience unacceptable toxicities and when continued treatment, is in the participant's best interest according to the Investigator.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals

ELIGIBILITY:
Inclusion Criteria:

• Participants enrolled into Part 1 must have tumor lesions where repeated IT injections are not feasible and in whom, based on the Investigator's judgement, SC injection is the only viable route of CMP-001 administration. Participants with lesions that are easily accessible for IT injections are not eligible to participate in Part 1. Participants enrolled into Part 2 must have at least one tumor lesion with a longest diameter of >/= 0.5 cm amenable for IT injection of CMP-001.

All participants enrolled into either Part 1 or Part 2 must meet all of the following inclusion criteria to be eligible:

* Histopathologically confirmed diagnosis of metastatic or unresectable malignant melanoma. Ocular melanoma participants are not eligible.
* Participants must have received prior treatment with anti-PD-1 or anti-PD-L1 therapy (alone or as part of a combination) in the advanced or metastatic setting and had documented progression per RECIST. Participants must have received at least 4 doses of anti-PD-1 or anti-PD-L1 therapy.
* Participants must have measurable disease by RECIST Version 1.1.
* Capable of understanding and complying with protocol requirements.
* A life expectancy of greater than 24 weeks at Screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Most recent laboratory values (within 3 weeks prior to Week 1 Day 1) meet the following standards:

  1. Bone marrow function: neutrophil count greater than or equal to (>/=) 1,000/cubic millimeter (mm^3), platelet count >/=75,000/mm^3 and hemoglobin concentration >/= 8.0 grams per deciliter (g/dL).
  2. Liver function: total bilirubin less than or equal to (<=) 1.5 times the upper limit of normal (ULN) of each institution, aspartate aminotransferase and alanine aminotransferase <=3 times the ULN range of each institution.
  3. Lactate dehydrogenase (LDH) <=2.0 times the ULN range of each institution.
  4. Renal function: serum creatinine <=1.5 times the ULN range of each institution.
* The participant must sign a written informed consent form prior to the initiation of any study procedures. Adult participants unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

* Pregnant or breast feeding
* Received investigational therapy (that is, small molecule or biologic) within 30 days prior to the start of CMP-001 dosing on Week 1 Day 1. However, if an investigational drug has a short half-life, a reduced wash out period may be acceptable upon permission given by the Sponsor.
* Received treatment with anti- cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody within 30 days prior to the start of CMP-001 dosing on Week 1 Day 1.
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Developed autoimmune disorders of Grade 4 while on prior immunotherapy. Participants who developed autoimmune disorders of Grade <=3 may enroll if the disorder has resolved to Grade <=1 and the participant has been off systemic steroids at doses greater than (>) 10 milligrams per day (mg/day) for at least 2 weeks.
* Require systemic pharmacologic doses of corticosteroids at or above the equivalent of 10 mg/day prednisone; replacement doses, topical, ophthalmologic and inhalational steroids are permitted. Participants who have a history of adrenal insufficiency and are receiving greater than 10 mg/day systemic steroids may be eligible but only after Sponsor consultation. Participants who are currently receiving steroids at a dose of <=10 mg/day do not need to discontinue steroids prior to enrollment.
* Active (that is, symptomatic or growing) central nervous system (CNS) metastases. Participants with CNS metastases are eligible for the trial if: a) the metastases have been treated by surgery and/or radiotherapy; b) the participant is off corticosteroids >10 mg/day and is neurologically stable for at least 2 weeks prior to Screening; c) brain MRI completed within 3 months of Screening.
* Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator, would make the participant unable to cooperate or participate in the trial.
* Severe uncontrolled cardiac disease within 6 months of screening, including but not limited to uncontrolled hypertension; unstable angina; myocardial infarction (MI) or cerebrovascular accident (CVA).
* Requires prohibited treatment that is, non-protocol specified anticancer. pharmacotherapy, surgery or conventional radiotherapy for treatment of malignant tumor)
* Women of child-bearing potential who are unable or unwilling to use an acceptable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Part 1: Dose-Escalation Phase: RP2D of CMP-001 When Administered SC and Given in Combination With Pembrolizumab | 15 days from date of first CMP-001 injection (Week 1 Day 1)
Part 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of CMP-001 (Week 1 Day 1) until 30 days after the last CMP-001 injection (up to approximately 2.5 years)
  TEAEs will be evaluated using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Part 1 Dose Escalation and Dose Expansion: Number of Participants With TEAEs | From first dose of CMP-001 (Week 1 Day 1) until 30 days after the last CMP-001 injection (up to approximately 2.5 years)
  TEAEs will be evaluated using CTCAE version 5.0.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Oral Temperature | From screening up to end of treatment (EOT) (up to approximately 2.5 years)
  Oral temperature should be measured in supine or seated position, following at least 30 minutes of rest.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Respiratory Rate | From screening up to EOT (up to approximately 2.5 years)
  Respiratory rate should be measured in supine or seated position, following at least 30 minutes of rest.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Systolic and Diastolic Blood Pressure | From screening up to EOT (up to approximately 2.5 years)
  Blood pressure should be measured in supine or seated position, following at least 30 minutes of rest.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Body Weight | From screening up to EOT (up to approximately 2.5 years)
  Physical examination included body weight measurement.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Body Mass Index (BMI) | From screening up to EOT (up to approximately 2.5 years)
  Physical examination included BMI measurement.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG) Parameters | From screening up to EOT (up to approximately 2.5 years)
  ECG parameters will include heart rate and PR, QRS, QT, and QT corrected for heart rate (QTc) intervals. QT will be corrected using Fridericia's (QTcF) formula. ECG will be performed after the participant has been resting in supine or semi-supine position for at least 5 minutes.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters | From screening up to EOT (up to approximately 2.5 years)
  Clinical laboratory parameters includes serum chemistry, hematology, urinalysis, coagulation and thyroid function tests.
Part 1 Dose Escalation: Concentration of Chemokine IP-10 | Day 1 of Weeks 1, 3, 15 and Day 2 of Week 3, 15
Part 1 and Part 2: Objective Response Rate (ORR) (Percentage of Participants With Objective Response) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Using Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) Scans | Baseline until confirmed disease progression (CR or PR) or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 2.5 years)
  ORR will be calculated as the number of participants with a confirmed complete response (CR) or partial response (PR) divided by the number of participants dosed.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Best Overall Response (BOR) Rate (Percentage of Participants With Best Objective Response of CR or PR) as per RECIST Version 1.1 Using CT or MRI Scans | Baseline until confirmed disease progression (CR or PR) or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 2.5 years)
  BOR will be calculated as the number of participants with best response of CR or PR divided by the number of participants dosed.
Part 1 Dose Escalation and Dose Expansion, and Part 2: Time to Response (TTR) as per RECIST Version 1.1 Using CT or MRI Scans | From first dose of CMP-001 until disease progression or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 2.5 years)
Part 1 Dose Escalation and Dose Expansion, and Part 2: Duration of Response (DOR) as per RECIST Version 1.1 Using CT or MRI Scans | From the date of first confirmed CR or PR until the first date of recurrent or progressive disease (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 2.5 years)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Pittsburgh Medical Center - Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided